CLINICAL TRIAL: NCT02141321
Title: SUB LINGUAL MISOPROSTOL PRIOR TO IUD INSERTION IN WOMEN WITH ONLY PREVIOUS CESARIAN SECTION: A Randomized Controlled Trial
Brief Title: Sub Lingual Misoprostol Before IUD Insertion in Women With Only Previous Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Mohamed S. Sweed lecturer of Obstetrics & Gynecology AinShams University., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9010023
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: IUD Insertion
Keywords: IUD; Misoprostol; Rectal administration
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): Women will receive two sub lingual tablets each containing 200 micro gram misoprostol (Misotac), receiving a total dose of 400 micro grams. Two hour later, Cu T 380A IUD (PREGNA) will be inserted.
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Women will receive two sub lingual placebo tablets which will be similar in size, color, odor and shape to the misoprostol tablets. Two hour later, Cu T 380A IUD (PREGNA) will be inserted.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Misotac; Cytotec; Misotec; Prostaglandin E1 synthetic analogue
  Arms: Misoprostol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the work is to evaluate the efficacy of the sub lingual prostaglandin E1 synthetic analogue (misoprostol) before IUD insertion to facilitate the procedure in patients delivered before only by cesarean section.

DETAILED DESCRIPTION:
The study will be conducted at Ain Shams University Maternity Hospital. 124 women candidate for Cu T 380A IUD insertion will be enrolled in the study. Half of them will receive 400 micro gram of misoprostol (Sigma) sub lingually and the other half will receive the placebo two hours before IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Normal size uterus.
* Willing to participate.
* Candidate for IUD insertion.
* Delivered only by cesarean section.
* Last delivery is more than 40 days before participating in the study.

Exclusion Criteria:

* Previous vaginal delivery
* Signs of genital infection.
* Menopause.
* Body mass index (BMI) > 35 kg/m2.
* Contraindication to misoprostol.
* Copper allergy.
* Positive pregnancy test.
* Had a prior attempt for IUD insertion.
* Uterine anomalies.
* Uterine fibroid.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain | During the procedure
  The perception of pain and discomfort as described by the patient assessed by Visual Analogue Scale (VAS). The scale will be graded from 0 to 10, 0 representing no pain at all and 10 worst possible imaginable pain.

SECONDARY OUTCOMES:
Difficulty of Procedure | During the procedure
  The degree of difficulty of the IUD insertion judged by the investigator as the resistance met at the internal cervical os. The procedure either graded as (easy), (moderate difficulty) or (difficult) or (failed insertion).
Complications | During the procedure and the following 24 hours.
  Uterine perforation, excessive bleeding, fever, IUD expulsion or any other unexpected complications will be assessed during the procedure and followed for the next 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Sweed, MD, Principal Investigator — Ain Shams University; Hassan A. Bayoumy, Professor, Study Director — Ain Shams University; Mohamed Y. Mohamed, M.B., B.Ch., Principal Investigator — Assiut University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt